CLINICAL TRIAL: NCT04628507
Title: Evaluation of Cell Free Preimplantation Genetic Testing
Brief Title: Cell Free Preimplantation Genetic Testing
Status: Not yet recruiting | Type: Observational
Sponsor: Genomic Prediction Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Genomic Prediction Inc 632
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Infertility, Female; Infertility, Male
Keywords: PGT; Noninvasive
MeSH Terms: conditions — Infertility, Female; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples, embryo spent culture medium, and leftover amplification product from embryo biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing IVF
  Interventions: Other: Spent media collection

INTERVENTIONS:
Other: Spent media collection — Embryo spent culture media, otherwise discarded as per standard of care, is collected once embryos have completed in vitro culture.

SUMMARY:
This study aims to develop preimplantation genetic testing methods from embryo culture media (cell free). Genetic testing of culture media will be compared to conventional methods based on embryo biopsies.

DETAILED DESCRIPTION:
Consenting patients will receive standard clinical IVF and PGT. Culture media from embryos will be collected for analysis. Collection of media will include laser assisted collapse of the blastocyst on day 5, 6, or 7 in order to release blastocoel fluid into the culture media. Embryos diagnosed as aneuploid or monogenic disorder affected (abnormal embryos) will be donated for additional analysis with patient consent.

Results obtained from culture media will not be provided to the patients. The information obtained from cf-PGT will be compared to results obtained from embryo biopsies obtained as part of routine PGT and evaluated for concordance and reliability. Abnormal embryos will be rebiopsied (~3 to 4 times) to evaluate concordance with cf-PGT and the original clinical trophectoderm biopsy PGT results.

All cases will be labelled using a 5-digit barcode and embryo number or saliva source code. Because PGT will be conducted under clinical regulatory approval (CAP and CLIA), patient information will be protected under HIPAA guidelines, including sending reports in encrypted secure email per standard operating procedures. All publications and presentations will maintain de-identification of any patient data used.

Patients may withdraw from the study at any time by contacting the principal investigator of their respective recruiting site. They will continue to receive standard of care through their treating IVF center. A recruitment target of 200 patients is intended for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF electing to utilize LifeView testing (PGT) will be offered participation in this study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing IVF electing to utilize LifeView testing who consented for embryo spent media collection and analysis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-06-11 (Estimated); Primary Completion 2027-11-11 (Estimated); Study Completion 2027-12-11 (Estimated)

PRIMARY OUTCOMES:
Concordance with PGT | 14 dyas
  Concordance rates with PGT diagnosis from trophectoderm biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Genomic Prediction Clinical Laboratory, North Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No